CLINICAL TRIAL: NCT00316160
Title: A Twelve-week, Multi-center, Randomized, Double-blind, Double-dummy, Parallel-group, Active Controlled, Escalating Dose Study to Compare the Effects on Sexual Functioning of Bupropion Hydrochloride Extended-release (WELLBUTRIN XL, 150-450 mg/Day) and Extended-release Venlafaxine (EFFEXOR XR, 75-225 mg/Day) in Subjects With Major Depressive Disorder
Brief Title: Sexual Functioning Study With Antidepressants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100368
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Depressive Disorder, Major; Major Depressive Disorder (MDD)
Keywords: sexual dysfunction; Depression; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Sexual Dysfunction, Physiological; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bupropion Hydrochloride Extended-release
Drug: Extended-release Venlafaxine
  Other Names: Bupropion Hydrochloride Extended-release

SUMMARY:
Effects of two depression medication on sexual functioning

DETAILED DESCRIPTION:
A Twelve-week, Multi-center, Randomized, Double-blind, Double-dummy, Parallel-group, Active controlled, Escalating Dose Study to Compare the Effects on Sexual Functioning of Bupropion Hydrochloride Extended-release (WELLBUTRIN XL, 150-450 mg/day) and Extended-release Venlafaxine (EFFEXOR XR, 75-225 mg/day) in Subjects with Major Depressive Disorder

ELIGIBILITY:
Inclusion criteria:

* Primary diagnosis of Major Depressive Disorder (MDD)
* must have met DSM-IV criteria for current major depressive episode for at least 8 weeks but no long than 2 years.
* HAM-D17 total score of >17 at screening and baseline.
* Severity of illness score of >4 at screening and baseline.
* Willing to discuss sexual functioning with investigator or designee.
* Sexual activity that leads to orgasm at least every 2 weeks.

Exclusion Criteria:

* Past or current DSM-IV diagnosis of Bipolar Disorder I or II, schizophrenia or another psychotic disorder(s).
* Primary DSM-IV diagnosis or received treatment for Panic Disorder, Obsessive Compulsive Disorder or Post Stress Disorder within previous 12 months.
* Poses a homicidal or serious suicidal risk, have made an attempt within months prior to screening or who has ever been homicidal.
* Myocardial infarction with 1 year of screening.
* Taken ibupropion hydrochloride or venlafaxine in the last 6 months.
* Positive urine test for illicit drug use or alcohol or substance abuse within the past 12 months.
* Psychotherapy within 3 months.
* Pregnant.
* Electroconvulsive therapy or transcranial magnetic stimulation within 6 months prior of screening.
* ECG or clinical evidence of atrial or ventricular hypertrophy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347
Dates: Start 2004-09; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
To compare the effects of bupropion XL and venlafaxine XR on overall sexual functioning in outpatients with MDD as measured by mean changes in CSFQ-S total scores across Weeks 5, 6, 9 and 12.

SECONDARY OUTCOMES:
Efficacy, Safety, Tolerability, Health Outcome

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (43):
- United States (43):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Temecula, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Coral Springs, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Smyrna, Georgia
  - GSK Investigational Site, Oak Brook, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Braintree, Massachusetts
  - GSK Investigational Site, Greenfield, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Lincoln, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Yakima, Washington
  - GSK Investigational Site, Middleton, Wisconsin

REFERENCES:
- [Result] Thase ME, Clayton AH, Haight BR, Thompson AH, Modell JG, Johnston JA. A double-blind comparison between bupropion XL and venlafaxine XR: sexual functioning, antidepressant efficacy, and tolerability. J Clin Psychopharmacol. 2006 Oct;26(5):482-8. doi: 10.1097/01.jcp.0000239790.83707.ab. PMID 16974189